CLINICAL TRIAL: NCT04424914
Title: GLOBAL PREVALENCE OF TRANSTHYRETIN AMYLOID CARDIOMYOPATHY (ATTR-CM) IN PARTICIPANTS WITH HEART FAILURE WITH PRESERVED EJECTION FRACTION (HFpEF)
Brief Title: Global Prevalence of ATTR-CM in Participants With HFpEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study early to not prolong timelines and to enable sharing of data collected which has potential to better support understanding of the prevalence of ATTR-CM in patients with HFpEF. Decision was not based on any safety findings.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B3461087; HFpEF ATTR-CM prevalence study (Other: Alias Study Number); 2020-002378-29 (EudraCT Number); ATTR-POP (Other: Alias Study Number)
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Transthyretin Amyloid Cardiomyopathy; Heart Failure With Preserved Ejection Fraction
Keywords: prevalence; transthyretin amyloid; ATTR-CM; HFpEF; scintigraphy
MeSH Terms: interventions — Radionuclide Imaging

STUDY DESIGN:
Intervention Model Description: To determine global prevalence of transthyretin amyloid cardiomyopathy in participants diagnosed with heart failure with preserved ejection fraction. No study treatment will be dispensed however, participants will undergo scintigraphy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATTR-CM positive (Other): Participants diagnosed with ATTR-CM by scintigraphy
  Interventions: Diagnostic Test: Scintigraphy
- ATTR-CM negative (Other): Participants who are scintigraphy negative for ATTR-CM
  Interventions: Diagnostic Test: Scintigraphy

INTERVENTIONS:
Diagnostic Test: Scintigraphy — scintigraphy

SUMMARY:
This study is a global, multi-center study designed to estimate the global prevalence of transthyretin amyloid cardiomyopathy (ATTR-CM) within a clinically at risk population [participants with heart failure with preserved ejection fraction (HFpEF)].

ELIGIBILITY:
Inclusion Criteria:

1. Medical history of heart failure (HF) with:

   1. At least 1 episode with clinical evidence of HF (without hospitalization) by signs or symptoms of volume overload or elevated intracardiac pressures that required/requires treatment with a diuretic for improvement; OR
   2. 1 prior hospitalization for HF.
2. Left ventricular ejection fraction (LVEF) >40%.
3. End-diastolic interventricular septal wall thickness (IVST) ≥12 mm.
4. Willing and able to undergo scintigraphy.

Exclusion Criteria:

1. Diagnosis of heart failure with reduced ejection fraction (HFrEF) (EF ≤40%).
2. Prior clinical history of myocardial infarction, CABG or multi-vessel obstructive coronary disease (>50% stenosis of ≥2 epicardial coronary arteries).
3. Presence or history of any severe valvular heart disease (obstructive or regurgitant).
4. A confirmed diagnosis of a non-amyloid infiltrative cardiomyopathy (ie, cardiac sarcoidosis, hemochromatosis), muscular dystrophies, cardiomyopathy with reversible causes, hypertrophic obstructive cardiomyopathy with known genetic etiology, or known pericardial constriction.
5. Any type of diagnosed amyloidosis (eg, amyloid A amyloidosis, primary [light chain] amyloidosis) or prior diagnosis of ATTR-CM.

   -

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (22):
  - Eastern shore Research Institute LLC, Fairhope, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Advance Medical Research Center, Miami, Florida
  - Bioclinical Research Alliance Inc., Miami, Florida
  - Biogenix Molecular, Miami, Florida
  - CIRA (Nuclear Imaging Facility), Miami, Florida
  - Nucleotron/ Doral Imaging Institute, CIRA DBA, Miami, Florida
  - Innova Pharma Research, Miami, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Stormont Vail Health, Topeka, Kansas
  - Cotton O'Neil Heart Center, Topeka, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Corewell Health, Grand Rapids, Michigan
  - Spectrum Health Medical Group Cardiovascular Medicine, Grand Rapids, Michigan
  - Cardiology Associates of North Mississippi, LLC, Tupelo, Mississippi
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - NYU Langone Health, New York, New York
  - WakeMed Health and Hospital, Raleigh, North Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - CardioVasc HR Inc, Saint-Jean-sur-Richelieu, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
- France (5):
  - Hôpital Louis Pradel, Bron
  - Centre Hospitalier Saint-Joseph Saint-Luc, Lyon
  - CHU Nimes - Hospital Caremeau, Nîmes
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse
  - Médecine Nucléaire de la Doua, Villeurbanne
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, BO
  - U.O. Clinica delle Malattie dell'Apparato Cardiovascolare - Ospedale Policlinico San Martino IRCCS, Genova, Genoa
  - U.O. Clinica delle Malattie dell'Apparato Cardiovascolare - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione IRCCS Policlinico San Matteo - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche, Pavia
  - Fondazione Toscana Gabriele Monasterio-UOC Cardiologia e Medicina Cardiovascolare, Pisa
- Japan (4):
  - Nagoya Tokushukai General Hospital, Kasugai, Aichi-ken
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Okayama University Hospital, Okayama
- Poland (4):
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - SPZOZ Uniwersytecki Szpital Kliniczny Im. Wojskowej Akademii Medycznej UM W Łodzi Centralny Szpital, Lodz, Łódź Voivodeship
- Spain (7):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari De Bellvitge, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
- St George's Hospital, St George's University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Yun S, Palladini G, Anderson LJ, Cariou E, Wang R, Angeli FS, Ebede B, Garcia-Pavia P. International prevalence of transthyretin amyloid cardiomyopathy in high-risk patients with heart failure and preserved or mildly reduced ejection fraction. Amyloid. 2024 Dec;31(4):291-301. doi: 10.1080/13506129.2024.2398446. Epub 2024 Sep 8. PMID 39245873
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461087

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 347 heart failure with preserved ejection fraction (HFpEF) participants within a clinically at-risk population were enrolled.
Groups:
- Participants With ATTR-CM: Participants enrolled in the study who were positive for transthyretin amyloid cardiomyopathy (ATTR-CM) by scintigraphy and were evaluable.
- Participants Without ATTR-CM: Participants enrolled in the study who were negative for ATTR-CM by scintigraphy and were evaluable.
- Non-evaluable Participants: Participants enrolled in the study who were non-evaluable.
Period: Overall Study
Arm/Group | Participants With ATTR-CM | Participants Without ATTR-CM | Non-evaluable Participants
Started | 56 | 259 | 32
Completed | 27 | 251 | 3
Not Completed | 29 | 8 | 29
Not completed — Other | 0 | 0 | 28
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Study terminated by sponsor | 23 | 7 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With ATTR-CM | Participants Without ATTR-CM | Non-evaluable Participants | Total
Number analyzed (Participants) | 56 | 259 | 32 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 84.13 (6.64) | 76.52 (7.87) | 75.56 (7.51) | 77.66 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 129 | 21 | 164
  Male | 42 | 130 | 11 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 99 | 9 | 130
  Not Hispanic or Latino | 33 | 158 | 23 | 214
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 20 | 1 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 11 | 6 | 23
  White | 48 | 226 | 25 | 299
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Global Prevalence of ATTR-CM in HFpEF Participants Clinically At-Risk of Disease Among Total Evaluable Participants
Description: Global prevalence of ATTR-CM in HFpEF participants was obtained by dividing the number of participants who were diagnosed with ATTR-CM in the study by the total number of HFpEF participants evaluated. Diagnosis of ATTR-CM was defined as: cardiac scintigraphy Grade 1, with confirmation of ATTR by cardiac biopsy; or cardiac scintigraphy Grade 2 or above. Exact 95% confidence intervals for the prevalence estimates were calculated using the method of Clopper and Pearson.
Time Frame: Day 1
Population: Evaluable analysis set included all participants who met the inclusion/exclusion criteria and completed Visit 1, excluding participants with cardiac scintigraphy assessed as non-evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Participants With HFpEF: All participants diagnosed with HFpEF who were noted with and without ATTR-CM.
Arm/Group | Participants With HFpEF
Number analyzed (Participants) | 315
Percentage of participants | 17.8 [13.72 to 22.46]

2. Secondary Outcome: Global Prevalence of ATTR-CM in Participants With HFpEF Clinically At-Risk of Disease by Subgroups (Regions, Age, Gender) Among Total Evaluable Participants
Description: The prevalence of ATTR-CM in HFpEF participants was evaluated for subgroups including regions (North America, Europe, and Asia), age categories (60-64 years, 65-69 years, 70-74 years, 75-79 years, 80-85 years, 85-89 years, >=90 years), and gender (male, female). The estimate of prevalence was defined as the number of participants meeting the diagnosis criteria of ATTR-CM divided by the number of evaluable participants in the study in the given subgroup category. Diagnosis of ATTR-CM was defined as: cardiac scintigraphy Grade 1, with confirmation of ATTR by cardiac biopsy; or cardiac scintigraphy Grade 2 or above. Exact 95% confidence intervals for the prevalence estimates were calculated using the method of Clopper and Pearson.
Time Frame: Day 1
Population: Evaluable analysis set included all participants who met the inclusion/exclusion criteria and completed Visit 1, excluding participants with cardiac scintigraphy assessed as non-evaluable. Here, "Number Analyzed" signifies number of participants evaluable for specified rows of the arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With HFpEF
Number analyzed (Participants) | 315
Percentage of participants
  Region: North America: number analyzed (Participants) | 83
  Region: North America | 4.82 [1.33 to 11.88]
  Region: Europe: number analyzed (Participants) | 210
  Region: Europe | 23.81 [18.22 to 30.16]
  Region: Asia: number analyzed (Participants) | 22
  Region: Asia | 9.09 [1.12 to 29.16]
  Age: 60-64 years: number analyzed (Participants) | 21
  Age: 60-64 years | 0 [0 to 0]
  Age: 65-69 years: number analyzed (Participants) | 34
  Age: 65-69 years | 5.88 [0.72 to 19.68]
  Age: 70-74 years: number analyzed (Participants) | 52
  Age: 70-74 years | 5.77 [1.21 to 15.95]
  Age: 75-79 years: number analyzed (Participants) | 68
  Age: 75-79 years | 14.71 [7.28 to 25.39]
  Age: 80-84 years: number analyzed (Participants) | 67
  Age: 80-84 years | 13.43 [6.33 to 23.97]
  Age: 85-89 years: number analyzed (Participants) | 54
  Age: 85-89 years | 44.44 [30.92 to 58.60]
  Age: >=90 years: number analyzed (Participants) | 19
  Age: >=90 years | 42.11 [20.25 to 66.50]
  Gender: Female: number analyzed (Participants) | 143
  Gender: Female | 9.79 [5.46 to 15.88]
  Gender: Male: number analyzed (Participants) | 172
  Gender: Male | 24.42 [18.20 to 31.54]

3. Secondary Outcome: Number of Participants According to TTR Genotypes Among Participants Diagnosed With ATTR-CM
Description: Number of participants diagnosed with ATTR-CM were evaluated for TTR genotypes (wild-type or hereditary form).
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Participants With ATTR-CM: Participants enrolled in the study who were positive for ATTR-CM by scintigraphy and were evaluable.
Arm/Group | Participants With ATTR-CM
Number analyzed (Participants) | 56
Participants
  TTR Genotype: Wild-Type | 47
  TTR Genotype: Variant | 7
  TTR Genotype: Not reported | 2

4. Secondary Outcome: Number of HFpEF Participants With and Without ATTR-CM Based on New York Heart Association (NYHA) Classification
Description: Participants were evaluated using the NYHA classification at Day 1. Class I: participants with cardiac disease but without resulting limitations of physical activity. Class II: participants with cardiac disease resulting in slight limitation of physical activity. Class III: participants with cardiac disease resulting in marked limitation of physical activity. Class IV: participants with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: Day 1
Population: Enrolled analysis set included all participants who met the inclusion/exclusion criteria and completed Visit 1.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With ATTR-CM: Participants enrolled in the study who were positive for ATTR-CM by scintigraphy.
- Participants Without ATTR-CM: Participants enrolled in the study who were negative for ATTR-CM by scintigraphy.
Arm/Group | Participants With ATTR-CM | Participants Without ATTR-CM
Number analyzed (Participants) | 56 | 259
Participants
  NYHA Classification: Class I | 2 | 26
  NYHA Classification: Class II | 43 | 165
  NYHA Classification: Class III | 8 | 66
  NYHA Classification: Class IV | 3 | 2
  NYHA Classification: Class I+II | 45 | 191
  NYHA Classification: Class III+IV | 11 | 68
Statistical Analysis 1: Comparison: Participants With ATTR-CM vs Participants Without ATTR-CM; Test type: Other; p = 0.3006, Chi-squared; p-values for comparison of proportions of CLASS I+II vs CLASS III+IV were based on a Chi-square test

5. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) in Participants With and Without ATTR-CM
Description: Participants were evaluated using NT-proBNP cardiac biomarker that was assessed at Day 1.
Time Frame: Day 1
Population: Enrolled analysis set included all participants who met the inclusion/exclusion criteria and completed Visit 1. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Nanogram per liter (ng/L)
Arm/Group | Participants With ATTR-CM | Participants Without ATTR-CM
Number analyzed (Participants) | 52 | 240
Nanogram per liter (ng/L) | 2470.0 [184.0 to 18449.0] | 817.5 [36.0 to 29370.0]
Statistical Analysis 1: Comparison: Participants With ATTR-CM vs Participants Without ATTR-CM; Test type: Other; p < 0.0001, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: Day 1 up to 6 months of follow-up
Arm/Group | Participants With ATTR-CM | Participants Without ATTR-CM | Non-evaluable Participants
All-Cause Mortality (participants affected / at risk) | 3/56 | 1/259 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/259 | 0/32
Other Adverse Events (participants affected / at risk) | 11/56 | 10/259 | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With ATTR-CM (N=56) | Participants Without ATTR-CM (N=259) | Non-evaluable Participants (N=32)
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Gravitational oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0 | 0
Posterior lens capsulotomy (Surgical and medical procedures) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04424914/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04424914/SAP_001.pdf